CLINICAL TRIAL: NCT03950947
Title: Effect of Permanent Internal Mammary Artery Occlusion on Extracardiac Coronary Collateral Supply: a Randomized Controlled Study
Brief Title: Effect of Permanent Right Internal Mammary Artery Occlusion on Extracardiac Coronary Collateral Supply
Acronym: IMAOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SNCTP000002493
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Circulation, Collateral; Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Ischemia
Keywords: Circulation, Collateral; Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional Study Arm (Experimental): In the presence of a significant right coronary artery stenosis and randomization to the intervention group, catheter-based occlusion of the right IMA distal to the take-off of the pericardio-phrenic branch is performed at baseline using a dedicated occlusion device (Amplatzer vascular plug, CE0086).
  Interventions: Device: Amplatzer vascular plug
- Sham-Control (Sham Comparator): In the presence of a significant right coronary artery stenosis, and randomization to the sham-procedure: right IMA will be selectively intubated using an appropriate catheter. Angiography of the RIMA and the pericardiacophrenic branch will be performed.
  Interventions: Other: Sham Controll

INTERVENTIONS:
Device: Amplatzer vascular plug — See above
  Arms: Interventional Study Arm
Other: Sham Controll — Angiography of the RIMA without occlusion
  Arms: Sham-Control

SUMMARY:
Coronary artery disease and the benefit of bypasses:

Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally, primarily consequence of myocardial infarction (MI). Coronary collaterals exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. Sufficient coronary collaterals have been shown to confer a significant benefit in terms of overall mortality and cardiovascular events. In this regard, the concept of augmenting coronary collateral function as an alternative treatment strategy to alter the course of CAD, as well as to control symptoms, is attractive.

Durable promotion of coronary collateral circulation:

Before the advent of coronary artery bypass grafting, permanent augmentation of coronary collateral supply by a single structural modification has already been attempted. Bilateral ligation of the internal mammary arteries (IMA) was performed in CAD patients to alleviate angina pectoris and electrocardiographic (ECG) signs of ischemia. The prevalent in vivo function of natural internal mammary arteries (IMA)-to-coronary artery bypasses and their anti-ischemic effect has been recently demonstrated by the investigators' research group. Levels of collateral function and myocardial ischemia were determined in a prospective, open-label clinical trial of permanent IMA device occlusion. In this study, coronary collateral function, has been shown to be augmented in the presence vs the absence of distal permanent ipsilateral IMA occlusion. These findings have been corroborated by the observed reduction in ischemia in the intracoronary ECG.

After this first step, the concept of permanent right IMA occlusion will be now investigated with a randomized, sham-controlled clinical trial.

DETAILED DESCRIPTION:
Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally. In industrialized countries, coronary artery disease (CAD) is the leading cause of death, consequence of myocardial infarction (MI).

In patients with acute coronary syndrome, percutaneous coronary intervention (PCI) has been shown to improve outcomes. For chronic stable CAD, a recent meta-analysis including more than 93'000 patients has concluded that there may be "evidence for improved survival with new generation drug eluting stents but no other percutaneous revascularization technology compared with medical treatment" . Conversely, a current review of recently published meta-analyses and the detailed analyses of 3 widely quoted individual studies indicate no difference exists among stable CAD patients between PCI and medical therapy regarding nonfatal myocardial infarct or all-cause or cardiovascular mortality. A very recently published randomized controlled trial among patients with stable, single-vessel CAD, the so called ORBITA trial, has found that PCI of the stenotic lesion did not prolong exercise time by more than the effect of a sham procedure during the short observation period of 6 weeks.

In contrast, coronary artery bypass grafting (CABG) was superior to PCI in patients with diabetes and multivessel CAD. CABG significantly reduced rates of death and myocardial infarction compared to PCI, but at a higher rate of stroke. Furthermore, in patients with advanced CAD, rates of myocardial infarction were more than 60% lower with CABG compared to PCI.

Conceptually, the benefit of CABG over PCI is not surprising as PCI targets significant coronary lesions thought to be responsible for causing ischemia. However, the deleterious effects of atherosclerosis are not typically preceded by significant luminal vascular narrowing. The vulnerable plaque eventually becoming the culprit plaque (causing myocardial infarction or sudden cardiac death) has typically a relatively mild stenosis. Furthermore, due to being multifocal and widespread, plaque vulnerability is not a target for, nor amenable to PCI.

Conversely, artificial - or natural - bypasses exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. Sufficient coronary collaterals have been shown to confer a significant benefit in terms of overall mortality and cardiovascular events.

In this regard, the concept of augmenting coronary collateral function (i.e. coronary arteriogenesis) as an alternative treatment strategy of revascularization to alter the course of CAD is attractive. In particular, promotion of natural coronary bypasses is an appealing concept for patients with CAD not or not entirely treatable by the conventional coronary revascularization methods of PCI and CABG. According to an analysis by Williams et al, 142 of 493 patients with chronic stable CAD (29%) belonged to the group with incomplete coronary revascularization (partial and no revascularization plus the so called no-option group), and this group showed reduced survival during the 3-year follow-up period. Coronary collateral function promotion from any source could, thus, contribute to the completeness of myocardial revascularization. Incomplete coronary revascularization in chronic CAD has been shown in a very large (n=35'993 patients), recently published registry-based study to reduce overall survival according to the number of vessels not treated by PCI and according to the severity of stenoses left untreated. Coronary arteriogenesis, i.e., the growth of pre-existing collateral vessels has to occur well in advance of acute atherothrombotic coronary artery occlusion in order to limit infarct size. The source of blood supply via natural coronary bypasses (collateral arteries) to a circulatory area at risk for infarction can be within the coronary circulation, but also via extracardiac paths, e.g., via internal mammary arteries (IMA; also termed internal thoracic arteries). Extracardiac coronary artery supply is conceptually related to the term coronary collateral circulation because of its known anatomical structure as arterial anastomoses between, e.g., IMA, the pericardium and coronary arterial branches. In an editorial, Kern and Seto recently commented the concept of "Stimulating extracardiac collaterals" as follows: "To be clinically relevant, coronary collaterals should be a sustainable and sufficiently large source of myocardial perfusion and reduce ischemia in daily life. It is conceivable that improved extracardiac collateral flow has the potential to be exactly that."

This study is relevant due to its primary clinical in addition to surrogate marker efficacy testing, which has not been performed so far for this new technique of coronary arteriogenesis. If proven useful to extend physical exercise time in the context of mitigated angina pectoris, a further option of myocardial revascularization for patients with CAD not treatable by PCI or surgical bypass or not rendered asymptomatic by medical therapy would be available. The catheter-based technique of IMA device occlusion is simple and safe, and if shown efficacious, its action would be potentially sustainable due to the durability of occlusion.

Preclinical Evidence:

The efficacy to augment blood flow via the IMA as naturally existing extracardiac bypasses has been shown in experimental studies in dogs. Bilateral IMA ligation has led to an acute average increase in total coronary flow of about 6-10 ml/min.

The prevalent in vivo function of natural IMA-to-coronary artery bypasses and their anti-ischemic effect has been recently demonstrated during temporary IMA balloon occlusion by the investigators' research group. 180 pairs of measurements were performed in 120 patients electively referred for coronary angiography. Levels of collateral function and myocardial ischemia were determined during two coronary balloon occlusions, the first with, the second without distal IMA balloon occlusion.

Coronary collateral function, as determined by collateral flow index (CFI) has been consistently increased in the presence vs the absence of distal ipsilateral IMA balloon occlusion. These findings have been corroborated by the observed reduction in ischemia as assessed by intracoronary ECG (icECG). Conversely, with distal contralateral IMA occlusion, collateral function and ECG signs of ischemia have remained unchanged.

Clinical Evidence to Date:

Surgical trials in humans on the effect of bilateral IMA ligation on angina pectoris were carried out in the late 1950ies among a total of close to 500 symptomatic CAD patients. Transthoracic access to the IMAs was performed under local anesthesia by a small incision between the 2nd and 3rd rib. The primary endpoint of the clinical trials was angina pectoris, and inconsistently, ECG signs of myocardial ischemia. While the uncontrolled trials reported favourable results in terms of symptomatic relief of angina pectoris, the subsequently performed sham-controlled, but very small trials of bilateral ligation showed similar improvement in the sham as in the verum group. A major limitation of these studies lies in the rather insensitive endpoints used, which preclude conclusions about the efficacy of IMA ligation on extracardiac coronary collateral function.

In a prospective, open-label proof-of-concept trial, the investigators' laboratory occluded the right IMA (RIMA) permanently using a 4-5mm vascular plug in 50 CAD patients. As primary study endpoint, CFI was obtained during ostial, 1-minute balloon occlusion of the untreated right coronary artery (RCA) at baseline before RIMA device occlusion and 6 weeks later. CFI changed from 0.071±0.082 at baseline to 0.132±0.117 (p<0.0001) at follow-up examination. The increase in RCA CFI was accompanied by a decrease in signs of myocardial ischemia during the brief coronary occlusion.

The acute functional changes observed by the investigators' study group in response to temporary distal IMA balloon occlusion as well as the improvement of collateral function in the right coronary artery with permanent distal IMA occlusion support the hypothesis that extracardiac coronary collateral supply can be augmented by this intervention.

However, the effect of permanent IMA occlusion was never investigated with a randomized clinical trial. Consequently, our study group conducts a study, whereby 100 patients with chronic stable CAD (single-blinded for the procedure) are randomly allocated (1:1) to the occlusion or to a sham control group. The study endpoints (CFI and icECG and clinical signs of myocardial ischemia during RCA occlusion) as well as the follow-up duration of 6 weeks are identical in the current and the previous proof-of-concept trial

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Referred for elective coronary angiography
* Written informed consent to participate in the study
* Significant stenosis of right coronary artery (FFR ≤0.80)

Exclusion Criteria:

* Acute coronary syndrome; unstable cardiopulmonary conditions, unstable angina pectoris
* Collateral flow index of right IMA <0.25
* Severe cardiac valve disease
* Congestive heart failure NYHA III-IV
* Prior coronary artery bypass surgery / prior cardiac surgery
* Coronary artery disease best treated by coronary artery bypass grafting
* Coronary artery disease unsuitable for intracoronary pressure measurements
* Prior Q-wave myocardial infarction in the vascular territory undergoing collateral function determination
* Severe renal or hepatic failure
* Women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in right coronary Collateral Flow Index (CFI) | Follow-up (week 6)
  Change from baseline in right coronary Collateral Flow Index (CFI) at follow-up (week 6) vs baseline

SECONDARY OUTCOMES:
Angina pectoris | Follow-up (week 6)
  Occurence of Angina pectoris during a controlled 1-minute ostial coronary occlusion for collateral flow index measurement. The occurence will be presented in percent (number of patient with Angina pectoris during occlusion / total number of patients * 100 ) per group (intervention and sham control). If no adequate collateral flow exists, all patient (=100%) should develop angina pectoris during a one-minute occlusion.
Change from baseline in intracoronary and surface ECG ST-segment shift during temporary right and left coronary balloon occlusion | Follow-up (week 6)
  Change from baseline in intracoronary and surface ECG ST-segment shift during temporary right and left coronary balloon occlusion at follow-up (week 6) vs baseline
Fractional Flow Reserve | Follow-up (week 6)
  Change in coronary FFR (unitless) at follow-up (week 6) vs baseline.
Number of patients with angiographic visibility of right IMA-to-coronary anastomoses | Follow-up (week 6)
  Angiographic visibility of right IMA-to-coronary anastomoses at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Seiler Christian, MD, Prof, Principal Investigator — Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stoller M, de Marchi SF, Seiler C. Function of natural internal mammary-to-coronary artery bypasses and its effect on myocardial ischemia. Circulation. 2014 Jun 24;129(25):2645-52. doi: 10.1161/CIRCULATIONAHA.114.008898. Epub 2014 Apr 17. PMID 24744276
- [Background] Moberg A. Anastomoses between extracardiac vessels and coronary arteries. II. Via internal mammary arteries. Post-mortem angiographic study. Acta Radiol Diagn (Stockh). 1967 May;6(3):263-72. doi: 10.1177/028418516700600306. No abstract available. PMID 6025072
- [Background] BLAIR CR, ROTH RF, ZINTEL HA. Measurement of coronary artery blood-flow following experimental ligation of the internal mammary artery. Ann Surg. 1960 Aug;152(2):325-9. doi: 10.1097/00000658-196008000-00018. No abstract available. PMID 13801236
- [Derived] Bigler MR, Stoller M, Tschannen C, Grossenbacher R, Seiler C. Effect of permanent right internal mammary artery occlusion on right coronary artery supply: A randomized placebo-controlled clinical trial. Am Heart J. 2020 Dec;230:1-12. doi: 10.1016/j.ahj.2020.09.006. Epub 2020 Sep 17. PMID 32949505